CLINICAL TRIAL: NCT00436540
Title: A Comparison Between Clobetasol Propionate (Clobex®) Spray and Clobetasol Propionate (Olux®) Foam With Regard to Efficacy, Safety, Preference and Duration of Response in Stable Plaque Psoriasis
Brief Title: A Comparison Between Clobetasol Propionate 0.05% (Clobex®) Spray and Clobetasol Propionate 0.05% (Olux®) Foam
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Ronald W. Gottschalk, MD / Medical Director, Galderma Laboratories, L.P.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: US10013
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2008-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Clobetasol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): clobetasol propionate (Clobex®) spray
  Interventions: Drug: Clobetasol Propionate 0.05% Spray
- 2 (Active Comparator): clobetasol propionate (Olux®) foam
  Interventions: Drug: Clobetasol Propionate 0.05% Foam

INTERVENTIONS:
Drug: Clobetasol Propionate 0.05% Spray — Apply to affected areas twice daily
  Other Names: Clobex® Spray
  Arms: 1
Drug: Clobetasol Propionate 0.05% Foam — Apply to affected areas twice daily
  Other Names: Olux® Foam
  Arms: 2

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of clobetasol propionate 0.05% (Clobex®) spray compared to clobetasol propionate 0.05% (Olux®) foam.

DETAILED DESCRIPTION:
Same as above.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a clinical diagnosis of moderate to severe plaque psoriasis, defined as 3%-20% of the body surface area involved

Exclusion Criteria:

* Subjects who have surface area involvement too large that would require more than 50 grams per week of Clobex® spray or more than 50 grams per week of Olux® foam
* Subjects whose psoriasis involves the scalp, face or groin
* Subjects with non-plaque psoriasis or other related diseases not classified as plaque psoriasis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2006-03; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Efficacy - Body Surface Area, Investigator Global Severity | 6 weeks

SECONDARY OUTCOMES:
Safety - Tolerability assessments, adverse events | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ronald W. Gottschalk, MD, Study Director — Galderma Laboratories, LP
Locations (2):
- United States (2):
  - Solano Clinical Research, Vallejo, California
  - Central Dermatology, PC, St Louis, Missouri